CLINICAL TRIAL: NCT02220049
Title: Phase I Dose Escalation of Velcade (Bortezomib) Daily Dose in Patients With Advances or Metastatic Solid Tumors
Brief Title: Dose Escalation of Velcade Daily Dose in Patients With Solid Tumors
Acronym: VELDAY
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Gustave Roussy, Cancer Campus, Grand Paris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2009-014354-15; 2009/1520 (Other: CSET number)
Record Dates: First submitted 2014-08-18; First posted 2014-08-19 (Estimated); Last update posted 2016-03-25 (Estimated); Status verified 2016-03

CONDITIONS: Advanced or Metastatic Solid Tumors
MeSH Terms: interventions — Bortezomib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Velcade (Experimental): Dose level Dose(mg/m²) d1-5, d8-12, d15-19 Cohort -2 Velcade 0.3 mg/m² Cohort -1 Velcade 0.4 mg/m² Cohort 1 Velcade 0.5 mg/m² Cohort 2 Velcade 0.6 mg/m² Cohort 3 Velcade 0.7 mg/m² Cohort 4 Velcade 0.8 mg/m² Cohort 5 Velcade 0.9 mg/m² Cohort 6 Velcade 1.0 mg/m² Cohort 7 Velcade 1.1 mg/m²
  Interventions: Drug: Bortezomib

INTERVENTIONS:
Drug: Bortezomib
  Other Names: VELCADE

SUMMARY:
VELCADE has demonstrated marked activity in haematological cancers leading to registration (MM, MCL).

Currently only biweekly or weekly regimens have been explored. Key signalling pathways which are aberrant in haematological cancers are also present in solid tumors.

VELCADE covers a broad spectrum of proteins, which are pivotal in carcinogenesis.VELCADE as a single agent & in combination with chemotherapy in solid cancers has shown modest and real anti-tumor activity but insufficient for Phase III development.

VELCADE PK exposure may be inadequate in solid tumors compared to "liquid cancers." VELCADE daily low dose administration may allow a greater PK exposure to be achieved, which is tolerated

Hypotheses:

VELCADE daily dosing (5-days on, 2-days off) is tolerable at biologically active doses VELCADE daily dosing (5-days on, 2-days off) results in increased PK (AUC)/PD (20S proteasome inhibition) VELCADE daily dosing (5-days on, 2-days off) with increased PK/PD results in improved anti-tumor activity (Increased tolerable VELCADE AUC may potentially cross the threshold required for clinically significant anti-tumor activity in solid cancers).

Some preclinical data suggest that: VELCADE daily dosing results in increased proteasome inhibition in tumor tissues Combination of VELCADE + XRT/other daily dosing agent may have increased anti-tumor activity compared to monotherapy alone.

ELIGIBILITY:
Inclusion Criteria:

1. Signed written informed consent
2. Target population

   * Subjects with advanced or metastatic solid tumors for whom the standard of care is ineffective or inappropriate
   * Ability to comply with visits/procedures required by the protocol
   * Life expectancy of at least 3 months
   * ECOG performance status score 0-1
   * Subjects with Histologic or cytologic diagnosis of any solid tumor (nonhematologic malignancy).
   * A tumor paraffin tissue block or 20-30 unstained slides from the tumor tissue block or enough slides from an FNA to allow for biomarker and predictive marker analyses. (This biopsy need not be obtained fresh at the time of screening. Obtaining unstained slides from the original diagnostic biopsy will suffice to meet this requirement).
   * Measurable or evaluable disease
   * Prior anti-cancer treatments are permitted (i.e. chemotherapy, radiotherapy, hormonal, or immunotherapy) with the following exceptions:
   * Toxicity related to prior therapy must either have resolved, returned to baseline or been deemed irreversible but does not conflict with exclusion criteria. Peripheral pre-existent neuropathy of any grade related or not related to previous anticancer therapy is an exclusion criterion.
   * At least 3 weeks must have elapsed since the last chemo-therapy, immunotherapy or radiotherapy and the beginning of protocol therapy. At least 6 weeks for nitrosoureas, mitomycin C and liposomal doxorubicin.
   * At least 3 weeks must have elapsed since the last anti-cancer hormonal therapy or antibody targeted therapy (e.g. Bevacizumab, Cetuximab, Trastuzumab). Hormonal treatment by analog LHRH will be allowed for patients with prostate cancer For extended-release formulations, the washout period must extend 1 month beyond the duration of activity of the formulation (e.g., 3 months for the activity of a depot formulation + 1 month wash out).
3. Age and Sex

   * men and women 18 - 75
   * Male and female patients of childbearing potential must use effective contraceptive measures during the study an d for at least 3 months after the end of the study treatment

Exclusion Criteria:

1. Sex and Reproductive Status

   * Male and female patients of childbearing potential who are unwilling or unable to use an acceptable method to avoid pregnancy for the entire study period and for up to three months after the study.
   * Male and female patients of childbearing potential using a prohibited contraceptive method.
   * Women who are pregnant or breastfeeding.
   * Women with a positive pregnancy test on enrollment or prior to study drug administration.
2. Target Disease Exclusions:

   Subjects who have documented unstable or untreated brain metastasis for at least 4 weeks and who are still requiring steroids (Subjects with treated and stably controlled CNS metastases for at least 4 weeks and are no longer on steroids are eligible for this study).
3. Medical History and Concurrent Diseases

   * A serious uncontrolled medical disorder or active infection, which would impair the ability of the subject to receive protocol therapy
   * History of thromboembolic disease or bleeding diatheses within the last six (6) months. This includes those subjects with tumors that were known to have spontaneously bled in the past.
   * History or presence of the diffuse interstitial lung disease or pericardial disease
   * Previous history or current presence of neurological disorders, including epilepsy, Parkinson's disease, multiple sclerosis, stroke.
   * Pre-existent peripheral neuropathy of any grade, related or unrelated to previous anticancer therapy. However, asymptomatic infraclinical neuropathy with moderate measurable changes revealed by EMG will be allowed.
   * Uncontrolled or significant cardiovascular disease including
   * myocardial infarction within 12 months- uncontrolled angina within 6 months
   * congestive heart failure within 6 months
   * LVEF ≤ 45% at baseline, or <55% if prior exposure to anthracyclines
   * diagnosed or suspected congenital long QT syndrome.
   * any history of clinically significant ventricular arrhythmias (such as ventricular tachycardia, ventricular fibrillation, or "Torsade de Pointes"). Controlled atrial fibrillation is not an exclusion criterion.
   * pericardial effusion
   * Subjects with concomitant other malignancies (except non-melanomatous skin cancers, early stage prostate or cervical cancers) are excluded unless a complete remission was achieved at least 5 years prior to study entry and no additional therapy is required or anticipated to be required during the study period
   * Subjects receiving any drugs or agents that inhibit (e.g., cimetidine, erythromycin, fluoxetine, ketoconazole, paroxetine) or induce (e.g., carbamazepine, glucocorticoids, phenobarbital, rifampin) CYP2C19 or CYP3A4 within 14 days before the first dose of VELCADE
   * Need for therapy with concomitant CYP 3A4 inhibitors (e.g., itraconazole,fluconazole,clarithromycin,erythromycin, norfloxacin, fluvoxamine, cimetidine, indinavir, ritonavir) or inducers (e.g., efavirenz, barbiturates, phenytoin, rifampin, glitazones)
   * Green tea consummation
4. Physical and Laboratory Test Findings (as confirmed by repeat test/results)

   * Inadequate bone marrow function defined as:
   * absolute neutrophil count < 1,500 cells/mm3.
   * platelet count < 100,000 cells/mm3.
   * hemoglobin < 9.0 g/dl
   * Inadequate hepatic function defined as:
   * total bilirubin > 1.5 times the institutional upper limit of normal (IULN) unless identified as a result of a confirmed genetic disorder of bilirubin metabolism (e.g., Gilbert's syndrome or familial benign unconjugated hyperbilirubinaemia).
   * alanine transaminase (ALT) and aspartate transaminase (AST) > 2.5 times the IULN
   * Inadequate renal function defined as serum creatinine >1.5 times the IULN
   * PT- INR/PTT >1.5 times the IULN is an exclusion criteria
   * If proteinuria ≥ 1+ then quantify by urinary protein in random urine sample; eligible if <1 g/l .
5. Allergies and Adverse Drug Reactions history of allergy to Velcade or chemically related compounds
6. Other Exclusion Criteria:

prisoners or subjects who are compulsorily detained (involuntarily incarcerated) for treatment of either a psychiatric or physical (e.g., infectious disease) illness must not be enrolled into this study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2010-12; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Identify maximum tolerated dose | Assessed every week from inclusion during the first 28 days and then every 28 days up to 19 months

SECONDARY OUTCOMES:
Efficacy | Assessed within 7 days of every cycle (28 days) up to 19 months
  According to the WHO criteria for tumor response

CONTACTS AND LOCATIONS:
Overall Officials: Rastislav BAHLEDA, MD, Principal Investigator — Gustave Roussy, Cancer Campus, Grand Paris
Locations (1):
- Gustave Roussy, Villejuif, Val de Marne, France